CLINICAL TRIAL: NCT03076216
Title: An Open Label, Single Arm Pilot Study of OncoSil™, Administered to Subjects With Unresectable Locally Advanced Pancreatic Adenocarcinoma, Given in Combination With Gemcitabine or Gemcitabine+Nab-paclitaxel Chemotherapies
Brief Title: A Pilot Study of OncoSil™ Given to Patients With Pancreatic Cancer Treated With Gemcitabine +/- Nab-paclitaxel.
Acronym: OncoPaC-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OncoSil Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC01P01
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2020-03

CONDITIONS: Unresectable Locally Advanced Pancreatic Carcinoma
Keywords: Pancreatic Cancer; Pancreas; metastases; pancreatic tumour; unresectable; locally advanced; implantable; radiographic; device; Phosphorous-32 (P32); OncoSil™; brachytherapy; gemcitabine; nab-paclitaxel; Abraxane
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- OncoSil™ plus SOC Chemotherapy (Other): OncoSil™ implanted with concurrent Standard of Care chemotherapy either gemcitabine or gemcitabine + Abraxane
  Interventions: Device: OncoSil™

INTERVENTIONS:
Device: OncoSil™ — The implantation of OncoSil™ under EUS

SUMMARY:
To evaluate the safety of OncoSil™ in a patient population undergoing standard chemotherapy treatment for pancreatic cancer. This study has been designed to satisfy FDA regulatory requirements.

The clinical investigation will be conducted at approximately 5 sites in the United States involving 20 patients.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate the safety of an active implantable (radiological) medical device OncoSil™, when implanted into patients with pancreatic cancer, in conjunction with Standard chemotherapy. OncoSil™, is an experimental treatment and carries the active treatment "radioactive Phosphorous (32P)" inside inactive silicon particles. Once implanted, the OncoSil™ Microparticles will stay in the tumour permanently. The purpose of OncoSil™, is to deliver the action of 32P directly into a targeted tumour to destroy cancer cells.

20 Patients will be taking part in a single arm open label research study - which means that everyone in the research study will receive the investigational treatment OncoSil™, plus their prescribed standard chemotherapy regimen which will be either Gemcitabine or Gemcitabine + nab-paclitaxel (Abraxane).

Endpoints: Primary Endpoint:

• Safety and Tolerability

Secondary Endpoints:

Efficacy

* Local Progression Free Survival (LPFS), within the pancreas
* Progression Free Survival (PFS), all sites
* Overall Survival (OS)
* Body weight
* Impaired function
* Pain Scores

The screening period will be performed within a 2 week period, followed by a treatment period of investigational visits which will occur weekly from Day 0 (Visit 1) until week 12, then 4 weeks later at week 16, and then at 8-weekly intervals until study participants reach documented progression of disease criteria for both LPFS and PFS which marks the end of study participation i.e. EOS visit.

8 weekly telephone contact will be used to monitor device or late radiation related adverse events, and oncology treatments/procedures administered for up to 12 months post OncoSil™ implantation. Overall survival will be conducted via 8 weekly medical record reviews and or telephone contact until subject death, or until 104 weeks post the last subject enrolled.

Overall survival will be conducted via 8-weekly medical record reviews until study participant death, or until 104 weeks post the last study participant enrolled.

Activity (Dose): The intended average absorbed radiation dose per treated tumour is 100 Gy (+20%).

Risks associated with OncoSil™ and/or implantation procedure

The following adverse events, considered to have a causal relationship with OncoSil™ or procedure, were recorded during previous clinical studies:

* Procedure-related pain
* Abdominal pain and discomfort
* Lethargy
* Fever
* Nausea and vomiting
* Abnormal liver function tests

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven adenocarcinoma of the pancreas.
2. Stage III unresectable locally advanced pancreatic carcinoma. Patients with technically resectable tumors (T1-T3) will also be eligible, if they are deemed unresectable due to medical comorbidities or refusal of surgery.
3. Pancreatic target tumor diameter of ≥ 2.0 cm (shortest axis) to ≤ 6.0 cm (longest axis), as qualified by the central reading center.
4. An ECOG Performance Status of 0 to 1 and Karnofsky Performance Status of 80 - 100.
5. Study participants' ≥ 18 years of age at screening.
6. To commence first-line standard gemcitabine and nab-paclitaxel chemotherapy, or gemcitabine alone, (per standard of care (SoC) according to the approved prescribing schedule), within 14 days post enrollment, with OncoSil™ implantation to occur during the fourth (4th) week of the first chemotherapy cycle.
7. Provide signed Informed Consent.
8. Willing and able to complete study procedures within the study timelines.
9. Adequate renal function: serum creatinine less than 1.5 x upper limit of normal (ULN).
10. Adequate liver function: serum liver transaminases ≤ 3 × ULN and serum bilirubin ≤ 1.5 × ULN*.

    * For study participants with recent biliary obstruction treated by drainage (e.g. stent), serum bilirubin of > 1.5 x ULN will be accepted for study entry provided that serial levels demonstrate clear improvement. In addition, chemotherapy should not be commenced until serum bilirubin is ≤ 1.5 × ULN.
11. Adequate bone marrow function: white blood cells (WBCs) ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1,500/mm3, hemoglobin ≥ 9 g/dL, and platelets ≥ 100,000/mm3.
12. Life expectancy of at least 3 months at the time of screening as judged by the investigator.
13. Treated with or eligible to commence prophylactic treatment with a proton-pump inhibitor prior to implantation, and to continue to receive treatment for at least 6 months post implantation.
14. Not pregnant, and if of childbearing potential, agrees to use adequate birth control (hormonal or barrier method of birth control or abstinence) prior to study entry and during the study and agrees not to donate sperm or ova, for the duration of the study and 12 months post implantation of the investigational device.

    -

Exclusion Criteria:

1. Evidence of distant metastases, based on review of baseline CT scan, as determined by the central reading center.
2. More than one primary lesion.
3. Any prior radiotherapy or chemotherapy for pancreatic cancer.
4. Use of other investigational agent at the time of screening, or within 30 days or five half-lives of Screening Visit 1, whichever is longer.
5. Pregnant or lactating.
6. In the opinion of the investigator, EUS directed implantation posing undue study participant risk. This includes:

   * where previous EUS-FNA was considered technically too difficult to perform;
   * imaging demonstrates multiple collateral vessels surrounding or adjacent to the target tumor within the pancreas;
   * presence (or significant risk) of varices near to the target tumor. Note: The feasibility of implantation of the target tumor and assessment of risk can be conducted at any time between Screening Visit 1 and the implantation date. A study participant should be considered for withdrawal prior to and including at the time of OncoSil™ treatment, if any of the above risk features become apparent following study participant screening and/or enrolment.
7. History of malignancy, treated or untreated, within the past five years whether or not there is evidence of local recurrence or metastases, with the exception of basal cell carcinoma of the skin and cervical carcinoma in situ.
8. Evidence of radiographic invasion into stomach or duodenum (if not certain, confirmation must be obtained prior to enrolment).
9. A known history of hypersensitivity to silicon or phosphorous, or any of the OncoSil™ components.
10. Any other health condition that would preclude participation in the study in the judgement of the investigator.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-11-28 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Safety / Tolerability of Device as determined by the number of treatment emergent adverse events (TEAEs) evaluated according to CTCAE V4.0 | Collected from the of signed informed consent until patient death or 104 weeks post last patient enrollment date, whichever is sooner]
  as determined by the number of treatment emergent adverse events (TEAEs) evaluated according to CTCAE V4.0

SECONDARY OUTCOMES:
Local Progression free survival within the pancreas | Assessed from Baseline through to first confirmed CT documentation of local progression within the pancreas, an average of 12 months
  As assessed by the central reader review of successive CT scans throughout the study
Progression free survival - entire body | Assessed from Baseline through to EOS visit - an average of 12 months
  As assessed by the central reader review of successive CT scans throughout the study
Overall survival | Assessed from Baseline to 104 weeks post last patient first study visit]
  As assessed by the time from participant consent to participant death or their survival to 104 weeks past the first study visit on the last subject enrolled in the study.
Body weight | Assessed from Baseline through to EOS visit, an average of 12 months
  Measurement of subject body weight at each study visit
Impaired function | Measured at each study visit for the duration of the study, an average of 12 months
  as measured by changes in the Karnofsky Performance Status from screening
Pain Scores | Measured at each study visit for the duration of the study, an average of 12 months
  Pain as measured by the numerical rating scale (NRS) at each study visit

OTHER OUTCOMES:
Tumor Response | Baseline measure from screening period, compared to Week 8 CT result, and then to 8 weekly CT results until local progression is determined, an average of 12 months
  as demonstrated by target tumour volumetric change (measured by a central reading centre)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M Herman, M.D., M.Sc., Principal Investigator — MD Anderson Cancer Centre
Locations (4):
- United States (4):
  - Cedars Sinai Department of Radiation Oncology, Los Angeles, California
  - Moffitt Cancer Centre, Tampa, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No